CLINICAL TRIAL: NCT05539547
Title: Effect of Neuromuscular Electrical Nerve Stimulation on Quadriceps Muscle Strength and Endurance in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effect of NMES on Quadriceps Muscle Strength and Endurance in Patients With COPD
Acronym: NMES
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Randall Debattista (Other)
Collaborators: University of Malta, Faculty of Health Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Randall Debattista, Master (By Research) Student, University of Malta
Organization: University of Malta (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FHS-2021-00004
Record Dates: First submitted 2022-09-04; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Chronic Obstructive Pulmonary Disease Moderate; Chronic Obstructive Pulmonary Disease Severe; Acute Exacerbation of COPD
Keywords: COPD; NMES; Quadriceps; Rectus Femoris; Strength; Endurance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Range of Motion, Articular

STUDY DESIGN:
Intervention Model Description: This study consists of the enrolment of two groups concurrently both receiving the usual physiotherapy treatment with the addition of NMES to the experimental group.
  Control Group: Effect of usual physiotherapy care, including chest and mobility physiotherapy on quadriceps strength and endurance during hospital admission on patients with severe acute exacerbation COPD.
  Experimental Group: Effect of NMES on quadriceps strength and endurance as an adjunct to usual physiotherapy care (chest physiotherapy and mobility) during hospital admission in patients with severe acute exacerbation COPD.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Sham Comparator): Patients shall receive the usual physiotherapy care, including chest and mobility physiotherapy on quadriceps strength and endurance during hospital admission on patients with severe acute exacerbation COPD.
  Interventions: Other: Usual Physiotherapy treatment (Chest Physiotherapy and mobility)
- Experimental Group (Experimental): Patients shall receive the investigated modality, NMES on quadriceps strength and endurance as an adjunct to usual physiotherapy care (chest physiotherapy and mobility) during hospital admission in patients with severe acute exacerbation COPD.
  Interventions: Device: Neuromuscular Electrical Nerve Stimulation

INTERVENTIONS:
Device: Neuromuscular Electrical Nerve Stimulation — Application of NMES on quadriceps muscle groups bilaterally
  Frequency: >50Hz Pulse duration: 350 - 400µs Intensity: Maximal tolerance (visible quadriceps muscle contraction and/or maximally tolerated by the patient, eliciting a slight discomfort) Time: 30 minutes per session, 7 sessions per week Duty Cycle: 2s on / 18s off Duration: Until discharge to a maximum of 30 days
  Arms: Experimental Group
Other: Usual Physiotherapy treatment (Chest Physiotherapy and mobility) — Daily chest physiotherapy and mobility
  Arms: Control Group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a respiratory condition that results in a mixture of small airway disease and parenchymal destruction, changes that are characteristic of emphysema. COPD is also characterized by persistent airflow limitation, an aspect which is noted to be a major cause of morbidity and disease burden worldwide. One in every 8 patients who suffer an exacerbation requires to be admitted to the hospital. Due to repercussions that arise both because of the systemic effects of COPD and also the aggravating factors due to the exacerbation, new adjuncts to treatment are being researched. NMES is a non-invasive and non-addictive means of muscle contraction and was introduced as a rehabilitation means post muscle injury, surgery, and eventually in certain diseases and its use in the treatment of patients with COPD is being looked into.

This research study shall adopt a quantitative approach. A Randomised Control Trial (RCT) shall be used to investigate the effect of Neuromuscular Electrical Nerve Stimulation on quadriceps muscle strength and endurance. Approximately 103 patients shall be randomly enrolled in the control group and the experimental group. The control group shall receive Physiotherapy as already provided by physiotherapists including chest and mobility exercises. The experimental group shall undergo Physiotherapy with the addition of NMES. To assess the effect of NMES on quadriceps strength and endurance, quadriceps strength shall be tested through the use of a hand-held dynamometer. Endurance shall be tested through a quadriceps endurance test which requires the leg to be extended against a weight corresponding to 70% of the 1 repetition maximum with a pace of 12 movements per minute, a test which will be stopped when the patient can no longer perform the movement despite strong verbal prompting and encouragement and the standardised 1-minute sit-to-stand. All tests are to be conducted before the intervention, hence on admission to the local general hospital and prior discharge to a maximum of 30 days from the date of admission. All tests shall be done in the patients' ward setting. Also, a diagnostic ultrasound scan of this group of muscles shall be performed upon admission and before discharge by a consultant radiologist at the radiology department. The Borg scale shall be used to assess the shortness of breath of the patients following the 1-minute sit-to-stand.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a respiratory condition that results in a mixture of small airway disease and parenchymal destruction, changes which are characteristic of emphysema. Research showed that COPD is also characterized by persistent airflow limitation, an aspect which some authors noted to be a major cause of morbidity and disease burden worldwide. One in every 8 patients who suffer an exacerbation of COPD requires to be admitted to the hospital. Literature also reported that re-admissions following discharge amounted to more than 20% within the first 20 days and continued to increase to approximately 33% within the first 90 days post-discharge from the hospital. Therefore, given that a high portion of patients will require further hospitalisations, this will impose a financial burden on the health care systems.

It emphasized the fact that apart from the pulmonary changes and respiratory impairments, patients diagnosed with COPD have systemic morphological and biomechanical changes. Morphological changes include a reduction in the cross-sectional area and a reduction in muscle mass. Biochemical changes are primarily due to long-term use of steroids and Chronic Systemic Inflammatory Syndrome (CSIS). Given such changes, more energy is required during activities of daily living (ADLs) by such patients, resulting in shortness of breath (SOB) following minimal exercises.

Due to muscle dysfunction, these patients develop physical deconditioning which is one of the primary symptoms reported. The primary cause of this relates to the ventilatory limitations present.

The severity of the condition and related pathophysiological changes also predict the level of exercise tolerance, with a worse condition resulting in increased levels of muscle atrophy, weakness affecting mostly the lower limbs, and poor oxidative capacity. In 2008, it was noted that the majority of patients with a severe form of COPD were so frail or dyspnoeic, making them unable to tolerate sufficient exercise training intensities required to improve their level of physical activity. Such patients were noted to become dyspnoeic following low-intensity physical activity, resulting in a decreased physical activity to control their SOB, with ultimately one-third of these patients exhibiting quadriceps muscle weakness related to immobility and decreased exercise tolerance.

Deterioration in muscle strength was the most commonly reported symptom characteristic of limb muscle dysfunction in people with COPD. In 2014, Mathur et al. noted that the occurrence of COPD patients experiencing early termination of exercise related to leg fatigue was approximately 40% more common than patients rating of SOB. A further 30% of the population sample reported equal leg fatigue and dyspnoea.

The higher the number of patients with COPD that become immobile, the more muscle mass is lost, and this loss continues to increase in periods of hospitalisation due to an exacerbation. Gosselink and Langer (2016) stated that immobility and inactivity both considerably contributed to muscle atrophy via the term "mechanical silencing".

Fear and immobility during and or exactly after an AECOPD also play a huge role in quadriceps strength. The deterioration in physical activity and muscle strength, primarily quadriceps muscle was noted throughout the course of the disease. It is further evident during the hospitalisation phase due to an acute onset of COPD.

Research has now changed its course of direction to find new methods and modalities which can assist COPD patients in maintaining some form of muscle activity even during their weakest days. Neuromuscular Electrical Nerve Stimulation (NMES) has been the most researched modality in combination with Pulmonary Rehabilitation (PR) with a variation in parameters use and duration of application.

NMES is a non-invasive means of muscle contraction and was introduced as a way for rehabilitation post muscle injury, surgery and eventually in certain diseases. NMES involves placing a conductive pad over the muscle and uses an intermittent electrical current to trigger action potentials and activate the intramuscular nerve branches and muscle fibres to generate a strong muscle contraction. It is a device which is self-administered, does not require supervision and carries a low metabolic load, providing an acceptable therapy for patients with a high symptom burden.

Therefore, after reviewing the above-mentioned gaps in literature where NMES is emerging as a promising modality in assisting patients with an exacerbating episode of COPD.

Methodology

To answer the research question stated above, a Randomised Control Trial (RCT) type of study design shall be adopted. An RCT is a study where participants are randomly assigned to an experimental and control group. As the study is conducted, the only expected difference between the control and experimental groups in a randomized controlled trial is the outcome variable being studied. This is important to approximate a controlled experiment, decrease bias and also improve statistical efficiency. In this research study, quadriceps strength, and endurance are the primary outcome variables. With the CAT and changes in rectus femoris, thickness and width through diagnostic ultrasound shall act as the secondary outcome measures.

Data collection shall focus on measuring quadriceps strength and assessing for structural changes, changes in the number of sit-to-stand repetitions for a duration of 1 minute and changes in the COPD Assessment Test (CAT) score. Patients shall be asked to carry out these tests on admission and on the same day of discharge from the hospital. A quantitative analysis will follow to determine whether NMES affected quadriceps muscle strength and endurance during an acute exacerbation of COPD. Concurrently, the same quantitative approach will be used to determine the severity of the patients admitted with an AECOPD to the hospital, alongside the level of anxiety and depression related to the chronic condition.

This research study will adopt a randomized-experimental research trial. Patients will be randomly assigned into two groups, the control group and the experimental group through an unpredicted randomised sequence and implementing the sequence that conceals the treatment until the patients are formally assigned to their groups. The control group shall receive the usual physiotherapy treatment currently offered to these patients in the ward setting by physiotherapists responsible for their care. Participants shall be given a unique code before the commencement of the study. All must have been previously diagnosed with COPD according to the Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) criteria which means that patients were presented with a Forced Expiratory Flow in one second (FEV1) of <70% of the predicted value and a Forced Expiratory Flow in one second to Forced Vital Capacity (FEV1: FVC) of <0.70.

Intervention

All patients enrolled will be randomly assigned into two groups, the control group and the experimental group. Every participant shall be given a code before the commencement of the study. The code will only be known to the researcher and the supervisor, the latter having no access to the computer used for data collection. The control group shall receive the usual physiotherapy treatment in their respective wards. The patients enrolled on the experimental group will have the usual physiotherapy treatment with the addition of NMES throughout their hospital stay. Electrodes shall be placed on the quadriceps group of muscles, bilaterally and concurrently.

Muscle stimulation is achieved using a portable stimulator, which can generate electrical pulses. The electrodes must be placed over the motor point of the muscle or muscle group to be stimulated. Amplitude, rate and waveform, which can also be referred to as the stimulus parameters, are adjusted to facilitate quality of movement and contraction without the muscle being fatigued throughout the treatment session (Hultman et al., 1983). NMES is described as an easy-to-use, easy-to-read and comfortable apparatus where the parameters are adjustable to the patient's progression, and programme recognition can be easily used by the patient.

These parameters have been chosen based on reports that concluded that a frequency of more than 50Hz stimulates cause a tetanic fusion, thus stimulating muscle contraction. Various other studies also supported such parameters

Ethical Considerations

Ethical approval was sought and approved by the University of Malta Research Ethics Committee (UREC). Patients will be instructed about the study through verbal and written information letters and consent will be requested. Informed consent will be needed from the participants and will be allowed to quit the research study when desired. All the data that will be collected regarding the patient will only be used for this study. All information gathered before and after the research study will be discarded upon completion.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the age of 40 - 79
2. Confirmed diagnosis of an Acute Exacerbation of COPD
3. MRC Dyspnoea score of 4 or above

Exclusion Criteria:

1. Any locomotor or neurological conditions
2. Malignancy or recent history of malignancy
3. Cardiac failure, pacemaker, and implantable cardioverter-defibrillator (ICD)
4. Distal arteriopathy, venous thromboembolism
5. Disabilities or recent orthopedic surgeries

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Quadriceps Strength | Week 0 and up to 30 days
  hand-held dynamometer shall be used to determine the muscle strength present before and after the intervention of the quadriceps muscle, irrespective of which group the patient is randomly enrolled to. Three readings shall be taken on each leg with the average recorded. Patients will sit at the edge of a bed, with the bed slightly elevated so that the lower limbs were in no time not in contact with the ground provided that the patient has sufficient static sitting balance.
Change in Quadriceps Endurance using the Quadriceps Endurance Testing | Week 0 and up to 30 days
  2. Quadriceps Endurance test: The quadriceps endurance test is performed with the patient sitting on a chair (White et a., 2013) with the starting position of 90 degrees knee and hip flexion with both arms crossed over the chest. The test consists of extending the dominant leg against weight corresponding to 70% of 1 repetition maximum with a pace of 12 movements per minute until exhaustion. The test shall stop when the participants could no longer follow the movements despite strong verbal prompting and encouragement. The duration is then recorded as the quadriceps endurance limit time (TlimQ, seconds).

SECONDARY OUTCOMES:
Change in 1 Minute Sit-to-stand | Week 0 and up to 30 days
  The 1 Minute Sit-to-Stand (1STST) is a well tolerable, sensitive, and reproducible test in COPD patients (Briand, J., 2018). This test is performed according to the American Thoracic Society guidelines (2002). Each participant is instructed to perform as much as tolerated sit-to-stands from a standardised 46cm height chair. The chair used shall have no arms and must rest against a wall. Patients shall be sitting upright on the chair, with knees and hips flexed at 90°, feet hip-width apart resting on the ground. Arms are held stationary by placing the hands on their hips. Patients are asked to indicate the level of dyspnoea and fatigue at rest. The Borg Dyspnoea Scale (0-10) hereunder explained is used. The number of repetitions of standing upright and then sitting down in the same position at a self-paced speed is counted for a duration of 1 minute. Participants are permitted to rest during the 1-minute duration while the time keeps on going.
Change in COPD Assessment Test Score (CAT Score) | Week 0 and up to 30 days
  The COPD Assessment Test Score, CAT Score is an eight-question questionnaire that will help both the patient-participant and also the healthcare professional to measure the symptoms and impact that COPD (Chronic Obstructive Pulmonary Disease) has on patient's wellbeing and daily life. The score was calculated on admission and prior discharge in-order to establish the effect NMES had on severe COPD patients.
Change in the Medical Research Council (MRC) dyspnoea scale | Week 0 and up to 30 days
  This scale was the main score used to stratify the severity of dyspnoea in respiratory disease, COPD during this study. The MRC is a scale ranging from 0 to 5 through which participants are allowed to specify the degree to which breathlessness is affecting their mobility. The five statements in the MRC dyspnoea scale describe the way patients perceive their dyspnoeic feeling.
Change in the Dyspnoea Breathlessness scale (Borg Dyspnoea Scale) | Week 0 and up to 30 days
  The Borg dyspnoea scale was carried out before and after the completion of the 1-Minute sit-to-stand test. The scale consists of numbers 0 to 10, where at number 0 patient's breathing is causing the patient no difficulty at all and progresses through to number 10 where the breathing difficulty is maximal. Patients enrolled in the study were instructed to indicate which number from the scale characterises the intensity of their breathlessness at that particular point in time. Prior to the 1-Minute sit-to-stand, participants were instructed to rate the effort of breathing, solely with no other experienced sensations.
Change in quadriceps muscle length and width | Week 0 and up to 30 days
  The rectus femoris muscle was identified and the thickness and width were measured pre and post-NMES intervention. The area for diagnostic ultrasound used was midway between the patellar tendon and the anterior superior iliac spine. Ramirez-Fuentes et al., (2018) assessed rectus femoris muscle using ultrasound in COPD patients during rehabilitation. They aimed to notice any correlation of muscle size with quadriceps strength and fat-free mass. Through their investigation, the muscle thickness was measured as the distance between deep and superficial aponeurosis. The width was calculated using the distance between the medial and lateral border of the muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tonio Agius, Physiotherapist, Study Chair — University of Malta, Faculty of Health Sciences